CLINICAL TRIAL: NCT00000597
Title: Multi-Center Trial of Anti-Thymocyte Globulin in Treatment of Aplastic Anemia and Other Hematologic Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 403
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2000-05

CONDITIONS: Anemia, Aplastic; Hematologic Diseases; Pancytopenia; Blood Disease
MeSH Terms: conditions — Anemia, Aplastic; Hematologic Diseases; Pancytopenia | interventions — Antilymphocyte Serum; Nandrolone

INTERVENTIONS:
Drug: antilymphocyte serum
Drug: nandrolone

SUMMARY:
To determine the therapeutic effects of anti-thymocyte globulin (ATG) in patients with aplastic anemia and related bone marrow failure diseases.

DETAILED DESCRIPTION:
BACKGROUND:

Aplastic anemia has been shown to respond to ATG. An immunological basis for aplastic anemia has been suggested by previous observations although the precise mechanism of action of ATG has not been defined. This serum, produced by immunization of horses with human thymocytes, may have broad reactivity with many human cells.

DESIGN NARRATIVE:

Patients in Group I with acute severe disease were randomized to receive ATG in either ten day or twenty-eight day courses. Patients in Group II with moderate or chronic disease were randomized to receive either ATG for ten days or high doses of the androgen, nandrolone decanoate. Patients in Group III with a variety of bone marrow diseases were also treated with ATG.

The study completion date listed in this record was inferred from the last publication listed in the Citations section of this study record.

ELIGIBILITY:
Men and women with moderate or acute, severe, aplastic anemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1982-03; Study Completion 1988-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Young — Laboratory of Hematology, NHLBI

REFERENCES:
- [Background] Young N, Griffith P, Brittain E, Elfenbein G, Gardner F, Huang A, Harmon D, Hewlett J, Fay J, Mangan K, et al. A multicenter trial of antithymocyte globulin in aplastic anemia and related diseases. Blood. 1988 Dec;72(6):1861-9. PMID 3058228